CLINICAL TRIAL: NCT06796153
Title: Assessment of the Protective Effect of Different Topical Agents on Visible Light Induced Pigmentation Compared with a Not Treated Control Zone
Brief Title: Photoprotection Efficacy of Different Topical Agents Under Visible Light Exposure
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: ACR_VLSP_21-02775
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Visible Light Exposure on Healthy Back Skin
Keywords: Photoprotection; Sunscreen; Visible Light (VL); Pigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Product 1: The test product 1 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 2: The test product 2 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 3: The test product 3 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 4: The test product 4 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 5: The test product 5 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 6: The test product 6 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 7: The test product 7 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Untreated zone: non-treated control zone
  Interventions: Other: Visible Light Exposure - Untreated zone

INTERVENTIONS:
Other: Visible Light Exposure - Treated zones — The treated zones were exposed to Visible Light to induce skin pigmentation (144J/cm2), 15 to 30 minutes after application.
  Groups: Product 1; Product 2; Product 3; Product 4; Product 5; Product 6; Product 7
Other: Visible Light Exposure - Untreated zone — The untreated zone was exposed to Visible Light to induce skin pigmentation (144J/cm2), as the same time as the treated zones.
  Groups: Untreated zone

SUMMARY:
To evaluate the protective effect of seven sunscreens on the pigmentation induced by visible light in comparison to an untreated control zone in healthy volunteers

DETAILED DESCRIPTION:
The sunscreens usually used as photoprotectors are known to protect in the UV domain (UVB and UVA). However, until recently visible light (400-700 nm) was considered as devoid of any photobiological effects on cutaneous tissue. Over the last two decades, with the development of photodynamic therapies and various dermatological treatments using visible laser light, several studies have reconsidered the cutaneous effect of visible light on the skin, in particular the induction of pigmentation.

The study intends to evaluate and to compare with a non-treated control zone and between them, the efficacy of photoprotective effect of different products after visible light exposure, between [400-700nm].

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female or male volunteer from 18 to 50 years old
2. Skin type III-IV according to the Fitzpatrick classification
3. Average ITA° (Individual Typologic Angle calculated value) on the back between 18° and 32° at screening and inclusion visits with an allowed difference of ± 2° between screening and inclusion visits
4. Uniform skin color over the eight zones (difference in ITA° between each zone should not be more than 4°)
5. Absence of freckles, naevi, hypo or hyper pigmented regions, hairs and marks of bronzing on the investigational area on the back
6. Female subject of childbearing potential, who is not sexually active, or using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study or menopausal female (with absence of menstruations for less than one year) or post-menopausal female (with absence of menstruations for more than one year)

   *Effective contraceptive methods: sexually active female of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide, intravaginal device, intrauterine device (IUD), condom with spermicide
7. Female of childbearing potential or menopausal female (with absence of menstruations for less than one year) willing to undergo urine pregnancy test
8. Subject willing and able to fulfil the study requirements and schedule
9. Subject informed about the study objectives and procedures, and able to understand them
10. Subject who has given written informed consent

Exclusion Criteria:

1. Subject who is pregnant or lactating or who is planning to become pregnant during the study
2. Subject with BMI > 30
3. Having planned UV exposure of the investigational area (sunlight or sunbeds) throughout the study
4. Having used sunbeds or had excessive sun exposure of the investigational area within the 3 months before inclusion
5. Having sunburn (erythema) on the back
6. Having dermatological disorders affecting the investigational area (presence of naevi, freckles, excess hair or uneven skin tones, vitiligo, photo-dermatological problems
7. History of skin cancer
8. History of abnormal response to sun
9. Presence of recent suntan (according to Investigator opinion) or photo-test marks
10. History of allergy, hypersensitivity, or any serious reaction to any cosmetic product
11. Any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator
12. Having used within the month before inclusion any systemic medication for more than 5 consecutive days (e.g. steroidal and non-steroidal anti-inflammatory drugs, corticoids, insulin, antihistamines, antihypertensive, antibiotics such as quinolone, tetracycline, thiazides, fluoroquinolones)
13. Having used within the month before inclusion any medication known to cause abnormal responses to UV exposure (e.g. vitamin A derivative, psoralen, aminolevulinic acid derivatives, etc.), or having planned to use these medications during the study
14. Having used within the 3 months before inclusion any depigmenting / whitening or pro-pigmenting topical treatments, or any systemic treatment that would interfere with the study assessments (anti-inflammatory drugs, corticoids, retinoids, hydroquinone, etc.) or having planned to use these treatments during the study
15. Having used, within the past 6 months, any physical treatment including laser or phototherapy (PUVA, IPL, PDT…) on the investigational area, or having planned to use these treatments during the study
16. Having planned to perform intensive sport (> 5 hours per week) or swim during the study
17. Subject who declares to be deprived of freedom by administrative or legal decision
18. Subject who cannot be contacted by telephone in case of emergency
19. Subject having participated within the 30 days before inclusion or currently participating in another clinical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers from 18 to 50 years old with phototype III to IV according to the Fitzpatrick scale and with an ITA° between 18° to 32° at Screening
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Pigmentation (Delta E - calculated values)

SECONDARY OUTCOMES:
Clinical investigator's assessment by using clinical scale | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Visual scoring of pigmentation, using a pigmentation 14-point scale with 0 (Absence), 1 (Barely visible), 2 (Very pale brown -), 3 (Very pale brown), 4 (Very pale brown +), 5 (Pale brown -), 6 (Pale brown), 7 (Pale brown +), 8 (Brown -), 9 (Brown), 10 (Brown +), 11 (Pronouced brown -), 12 (Pronouced brown), 13 (Pronouced brown +) Visual scoring of erythema, using an erythema 14-point scale with 0 ((Absence), 1 (Barely visible), 2 (Very pale pink -), 3 (Very pale pink), 4 (Very pale pink +), 5 (Pale pink -), 6 (Pale pink), 7 (Pale pink +), 8 (Pink -), 9 (Pink), 10 (Pink +), 11 (Pronouced pink -), 12 (Pronouced pink), 13 (Pronouced pink +)
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Pigmentation : Individual Typologic Angle (ITA° - calculated value) based on Delta L* and Delta b* - calculated values)
Safety / Local Tolerance | From the informed consent signature date until the end of the study (Day 5)
  Safety was assessed by recording Adverse Events, including cutaneous reactions (local intolerance).
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure)
  Erythema (Delta a* - calculated value)

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Biotechnology S.R.L, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No